CLINICAL TRIAL: NCT04497688
Title: A Multi-center, Open-label, Single-arm Study to Evaluate the Efficacy and Safety of PEG-rhG-CSF(Jinyouli®) in Preventing Neutropenia After Chemotherapy in Patients With Non-Hodgkin's Lymphoma
Brief Title: Evaluate the Efficacy and Safety of PEG-rhG-CSF in Preventing Neutropenia After Chemotherapy in Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC -JYL-NHL-03
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Non Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEG-rhG-CSF group (Experimental): Patients received subcutaneous injection of PEG-rhG-CSF(Jinyouli®) 48 hours after the end of chemotherapy, 6mg for patients with body weight≥45kg and 3mg for patients with body weight less than 45kg, once per chemotherapy cycle
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — Patients received a single dose of PEG-rhG-CSF per cycle. The chemotherapy regimen must meet the interval between two chemotherapy sessions at least 12 days.

SUMMARY:
The main treatments for non-Hodgkin's lymphoma are surgery, radiotherapy, chemotherapy, and bone marrow transplantation. Neutropenia is the most common and serious complication of most chemotherapy. This study is a multi-center, open-label, single-arm clinical study to evaluate the efficacy and safety of jinyouli in preventing neutropenia in patients with non Hodgkin's lymphoma after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, gender is not limited;
2. Patients with lymphoma diagnosed by histopathology or cytology;
3. Patients requiring multi-cycle chemotherapy;
4. Planned chemotherapy regimen FN risk ≥ 20 % , or 10% <FN risk < 20% with high risk factors ; According to the judgment of the investigator, there is a risk of FN occurrence if G-CSF support is not accepted, PEG-rhG-CSF should be used prophylactically from the first cycle;
5. Physical status (KPS) score ≥ 70 points;
6. Expected Survival period of more than 3 months;
7. Normal bone marrow hematopoietic function (ANC ≥1.5×10^9/L, PLT≥80×10^9/L, Hb≥75g/L, WBC≥3.0×10^9/L);
8. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5 times the upper limit of normal value, or≤5 times the upper limit of normal value when there is liver metastasis; total bilirubin (TBIL)≤2.5 times the upper limit of normal value; serum creatinine (Cr)≤2 times the upper limit of normal value;
9. Female patients of childbearing age must be negative in urine pregnancy test before treatment;
10. The testers (or their legal representatives/guardians) must sign an informed consent form.

Exclusion Criteria:

1. Lymphoma central involvement;
2. Hematopoietic stem cell transplantation or organ transplantation;
3. Local or systemic infection without adequate control;
4. Severe internal organ dysfunction and occurred in the last 6 months Myocardial infarction;
5. Those who used other test drugs of the same kind or accepted other clinical trials within 4 weeks before enrollmen；
6. Allergy to PEG-rhG-CSF, rhG-CSF and other preparations or proteins expressed by Escherichia coli;
7. Severe mental illness, affecting informed consent and/or adverse reaction expression or observation;
8. Pregnant or lactating female patients; women who refuse to accept contraceptive measures ;
9. Researchers determine unsuited to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade Ⅲ/Ⅳ neutropenia | From date of randomization until the date of the study completion，up to 24 weeks
  Grade Ⅲ neutropenia is defined as ANC≥0.5×10^9/L, and <1×10^9/L; Grade Ⅳ neutropenia is defined as ANC<0.5×10^9/L

SECONDARY OUTCOMES:
Incidence of febrile neutropenia (FN) | From date of randomization until the date of the study completion，up to 24 weeks
  A single oral temperature is 38.3℃ or ≥38℃ for more than 1 h, and the absolute value of neutrophils is less than 0.5×10^9/L or the absolute value of neutrophils is less than 1.0×10^9/L but it is expected to drop to less than 0.5×10^9/L within 48 hours
Antibiotic use rate | From date of randomization until the date of the study completion，up to 24 weeks
  Antibiotic use rate during the treatment cycle
Incidence of dose adjustment of chemotherapy or delay of chemotherapy | From date of randomization until the date of the study completion，up to 24 weeks
  Dose adjustment is defined as the reduction of planned dose of chemotherapy; Chemotherapy delay is defined as the delay in starting the next planned chemotherapy for more than 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Lihong Liu, PHD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- The fourth hospital of Hebei Medical University, Shijiazhuang, Hebei, China